CLINICAL TRIAL: NCT07177677
Title: Intravenous Injection of Human Bone Marrow Mesenchymal Stem Cell (hBMMSC) in the Treatment of Autism Spectrum Disorder (ASD): An Exploratory Study on the Safety and Preliminary Efficacy
Brief Title: A Study of Mesenchymal Stem Cell in the Treatment of Autism Spectrum Disorder
Acronym: ASD
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiuzhitang Maker (Beijing) Cell Technology Co.,Ltd. (Other)
Collaborators: Capital Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MKMSC-CT-003-1
Record Dates: First submitted 2025-09-02; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Autism Spectrum Disorder
Keywords: human Bone Marrow Mesenchymal Stem Cell (hBMMSC); Autism Spectrum Disorder (ASD)
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hBMMSC 0.5×10^6 cells/kg (Experimental): human Bone Marrow Mesenchymal Stem Cell (hBMMSC) 0.5×10^6 cells/kg、 1.0×10^6 cells/kg、 2.0×10^6 cells/kg
  Interventions: Biological: hBMMSC

INTERVENTIONS:
Biological: hBMMSC — Group 1: 0.5×10^6 cells/kg (participant's body weight) single dose; Group 2: 1.0×10^6 cells/kg (participant's body weight) single dose; Group 3: 2.0×10^6 cells/kg (participant's body weight) single dose.
  Other Names: human Bone Marrow Mesenchymal Stem Cell

SUMMARY:
This clinical trial aims to evaluate the safety and preliminary efficacy of intravenous administration of human bone marrow-derived mesenchymal stem cells (hBMMSCs) in patients with autism spectrum disorder (ASD).

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a neurodevelopmental disorder characterized primarily by impaired social communication, restricted interests, and repetitive, stereotyped behaviors. Currently, there are no effective therapeutic drugs, and main interventions consist of educational rehabilitation and behavioral management.The purpose of this study is to evaluate the safety and preliminary efficacy of hBMMSC intravenous treatment in patients with ASD. The clinical trial intends to involve 42 participants. The trial is expected to last approximately 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥6 years old
* Body weight ≥ 17 kg
* Meets the diagnostic criteria for Autism Spectrum Disorder (ASD) as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), and confirmed by the Autism Diagnostic Interview-Revised (ADI-R) and the Autism Diagnostic Observation Schedule-2 (ADOS-2)
* Has either not received any psychotropic medication in the three months prior to enrollment or has been on a stable regimen of psychotropic medication for at least three months
* The subject and/or their legal guardian(s) agree to participate in the trial and provide signed informed consent.

Exclusion Criteria:

* Inability of the subject or their guardian to sufficiently understand instructions in Chinese
* Active infection (viral, bacterial, fungal, or mycobacterial)
* A confirmed diagnosis of Rett syndrome, childhood disintegrative disorder, fragile X syndrome, or other genetic/metabolic diseases that may impact cognitive development
* History of epileptic seizures within 6 months prior to enrollment
* History of suicide attempts/self-harm, presentation of suicidal ideation, or being judged as the risk of suicidal by the investigator
* Severe hematologic diseases or active malignancy
* Severe hepatic or renal disease
* Participation in a drug clinical trial within 3 months prior to enrollment (unless beyond the protocol-defined wash-out period) or participation in any other stem cell study within the past year
* A positive skin test result
* Any other condition which, in the opinion of the investigator, would make the subject unsuitable for participation in this study

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Safety Evaluation of hBMMSC Injection in ASD Patients | 48 weeks
  Adverse events and serious adverse events.

SECONDARY OUTCOMES:
Preliminary Efficacy Evaluation of hBMMSC Injection for Patients with ASD | 48 weeks
  Changes in the scores of the Adaptive Behavior Assessment System (ABAS), Autism Behavior Checklist (ABC), Clinical Global Impression (CGI), Autism Treatment Evaluation Checklist (ATEC), Social Responsiveness Scale(SRS), Repetitive Behavior Scale-Revised (RBS-R), as well as the levels of blood inflammatory factors.

IPD SHARING:
Plan to Share IPD: No